CLINICAL TRIAL: NCT00912522
Title: Magnetic Prefrontal Stimulation for Studying the Role of the Cortex in High-level Cognition Processes and Reward System
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Moshe Isserles, MD, Hadassah Medical Organization
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 0116-09-HMO-CTIL
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Healthy Volunteers
Keywords: reward; TMS; cognition; Motivation; Perception; Decision making

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- LT PFC HIGH FREQ TMS (Active Comparator)
  Interventions: Device: TMS
- LT PFC LOW FREQ TMS (Active Comparator)
  Interventions: Device: TMS
- RT PFC HIGH FREQ TMS (Active Comparator)
  Interventions: Device: TMS
- RT PFC LOW FREQ TMS (Active Comparator)
  Interventions: Device: TMS
- SHAM STIMULATION (Sham Comparator)
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — TRANSCRANIAL MAGNETIC STIMULATION

SUMMARY:
The investigators intend to study the role of the cortex in high- level cognition processes and sensory adaptation, by the use of non-invasive Transcranial Magnetic stimulation and various cognitive tests.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women, age of 18-60
* answered negatively to questions of TMS safety questionnaire
* signed and declared about their agreement to participate in the study
* hebrew speaker

Exclusion Criteria:

* self history of significant mental disorder
* self history or first-degree relatives history of epilepsy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2009-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes in scoring of different tests and questionnaires | One year

SECONDARY OUTCOMES:
Correlation of different tests and questionnaires | One year

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Isserles, Dr., Principal Investigator — Hadassa Medical Organization
Locations (1):
- Hadassah medical org, Jerusalem, Israel